CLINICAL TRIAL: NCT04862676
Title: A Pilot Study to Determine the Safety and Efficacy of Repeated Hyperbaric Oxygen Therapy in Multiple Myeloma Patients Undergoing High-Dose Therapy and Autologous Stem/Progenitor Transplantation
Brief Title: Repeated HBO Therapy in Myeloma Patients Undergoing High-Dose Therapy and Auto-HCT
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Rochester (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Omar Aljitawi, Associate Professor of Hematology/Oncology, University of Rochester
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UMMY19160; R37CA225791 (NIH)
Record Dates: First submitted 2020-11-06; First posted 2021-04-28 (Actual); Last update posted 2025-09-10 (Actual); Status verified 2025-09

CONDITIONS: Myeloma
MeSH Terms: conditions — Neoplasms, Plasma Cell | interventions — Hyperbaric Oxygenation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Experimental Arm:single (Experimental): Repeated treatments with hyperbaric oxygen on Days 0, +1 and +2 of high-dose therapy melphalan and autologous transplants.
  Interventions: Drug: Hyperbaric oxygen

INTERVENTIONS:
Drug: Hyperbaric oxygen — The treatment consists of exposure to hyperbaric oxygen at 2.5 atmospheric absolutes (ATA) for a total of 90 minutes after compression to 2.5 atmosphere absolutes (ATA) in a monoplace hyperbaric chamber breathing 100% oxygen. The subjects will be in the chamber for a total of 120 minutes as approximately 10-15 minutes are spent during the compression and decompression phases and subjects have 5-10 minute room air breaks every 30 minutes of hyperbaric oxygen treatment.

SUMMARY:
Subjects with multiple myeloma (MM) who are considered eligible for high-dose therapy and autologous stem cell transplantation by the transplant team at WCI will be enrolled in the study.

DETAILED DESCRIPTION:
Subjects with multiple myeloma (MM) who are considered eligible for high-dose therapy and autologous stem cell transplantation by the transplant team at WCI will be enrolled in the study. Subjects will receive HBO therapy on Days 0, +1 and +2 of the transplant. The treatment consists of exposure to hyperbaric oxygen at 2.5 atmospheric absolutes for a total of 90 minutes after compression to 2.5 atmosphere absolutes in a monoplace hyperbaric chamber (Model 3200/3200R, Sechrist Industries, Inc., USA), breathing 100% oxygen. Subjects will be in the chamber for a total of 120 minutes as approximately 10-15 minutes will be spent during the compression and decompression phases and subjects will have 5-10 minute room air breaks every 30 minutes of hyperbaric oxygen treatment. Subjects will be seen daily until neutrophil recovery is documented . After neutrophil recovery is documented, the subjects will be seen in clinic at least weekly through day +100. A final visit will be scheduled day +100. As part of routine care, subjects will be followed daily or as directed by the treating physician until neutrophil recovery, defined as three consecutive days of achieving a neutrophil count of >500/mm3. Laboratory testing will occur per institutional guidelines. Follow-up will continue until Day +100. Donor chimerism and disease status will be determined by bone marrow biopsy on Day +30 and day +100 post-transplant.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with Multiple myeloma
* Subjects must be 18 years old
* Karnosfsky Performance of greater than 70 percent
* Adequate hepatic, cardiac and pulmonary function
* Subjects should have New York Heart Association Functional Classification of: Class 1 or Class II.

Exclusion Criteria:

* Pregnant or breastfeeding
* Severe chronic obstructive pulmonary disease requiring oxygen supplementation
* History of spontaneous pneumothorax
* Active ear/sinus infection
* Sinus surgery within the last 5 years
* Claustrophobia
* History of recurrent seizures within 5 years of study enrollment
* Evidence of pneumothorax or significant pulmonary fibrosis on chest imaging within 60 days of transplant
* Prior chest surgery involving thoracotomy or prior direct irradiation to the lungs
* Subjects who have had intrathecal chemotherapy within 2 weeks of starting preparative regimen or cranial irradiation within 4 weeks of starting preparative regimen
* Active and uncontrolled viral, fungal or bacterial infection
* Use of tobacco 72 hours prior to transplant

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2022-04-22 (Actual); Primary Completion 2025-04-04 (Actual); Study Completion 2025-06-30 (Actual)

PRIMARY OUTCOMES:
Number of participants with a treatment-limiting toxicity | 24 hours
  Treatment-limiting toxicities (defined as the occurrence of any of the following complications within 24 hours of HBO: Seizure disorder, pneumothorax, death, any irreversible grade Ill or any grade IV toxicity that is determined by the treating physician to be at least likely related to HBO therapy) will be assessed 24-hours post-hyperbaric oxygen therapy.
Number of participants with an AE or SAE attributed to HBO therapy. | 100 days
  Possible long-term effects of hyperbaric oxygen therapy treatment prior to autologous peripheral blood stem cell transplant will be assessed at day +100 post-transplant. AEs and SAEs will be graded using CTCAE version 5.

SECONDARY OUTCOMES:
Time to neutrophil recovery | 100 days
  Based on the patient having achieved three consecutive days of Absolute Neutrophil Count (ANC) ≥ 500/microliter

CONTACTS AND LOCATIONS:
Overall Officials: Omar Aljitawi, MMBS, Principal Investigator — University of Rochester
Locations (1):
- James P. Wilmot Cancer Center at University of Rochester Medical Center, Rochester, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
All individual data collected during the trial will be shared after deidentification, including dictionaries.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Data will be available immediately following publication. No end date.
Access Criteria: Anyone who wishes to access the date for any type of analyses.